CLINICAL TRIAL: NCT00729859
Title: Hormonal Regulation of Circulating Endothelial Progenitor Cells and HDL-C in Men Title Changed With New Protocol (12/14/09): Hormonal Regulation of HDL-C in Men
Brief Title: CEP-1 Hormonal Regulation of Circulating Endothelial Progenitor Cells and HDL-C in Men
Acronym: CEP-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Stephanie T. Page, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 33853-A; U54HD042454 (NIH)
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: HDL; Insulin sensitivity; testosterone; estradiol; cholesterol
MeSH Terms: conditions — Insulin Resistance | interventions — acyline; Anastrozole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Acyline 300 µg/kg injections every two weeks (2 doses) + placebo (no active ingredients) gel daily for 28 days + oral placebo pill daily for 28 days
  Interventions: Drug: Acyline
- Group 2 (Experimental): Acyline 300 µg/kg injections every two weeks (2 doses) + Testosterone gel 100 mg daily for 28 days + oral placebo pill daily for 28 days
  Interventions: Drug: Acyline + Testosterone gel
- Group 3 (Experimental): Acyline 300 μg/kg injections every two weeks (2 doses) for 28 days + Testosterone gel 100 mg daily for 28 days + oral anastrozole pill 1 mg daily for 28 days
  Interventions: Drug: Acyline + testosterone gel + anastrozole

INTERVENTIONS:
Drug: Acyline — Acyline 300 μg/kg injections every two weeks (2 doses) for 28 days + placebo Testosterone gel daily for 28 days + placebo oral anastrozole pill daily for 28 days
  Other Names: placebo testosterone gel; placebo pill
  Arms: Group 1
Drug: Acyline + Testosterone gel — Acyline 300 μg/kg injections every two weeks (2 doses) for 28 days + Testosterone gel 100 mg daily for 28 days + placebo oral pill 1 mg daily for 28 days
  Other Names: Acyline; testosterone gel
  Arms: Group 2
Drug: Acyline + testosterone gel + anastrozole — Acyline 300 μg/kg injections every two weeks (2 doses) for 28 days + Testosterone gel 100 mg daily for 28 days + oral anastrozole pill 1 mg daily for 28 days
  Other Names: Acyline; Testosterone gel; Anastrozole
  Arms: Group 3

SUMMARY:
The original purpose of this research study was to understand the effects of testosterone (T) and estrogen on stem cells in the blood. The knowledge would be used to help understand the effects of T and estrogen on cardiovascular (heart and blood vessel) disease, and to help in the development of a safe male hormonal contraceptive.

The effect of androgens on the number of circulating endothelial progenitor (CEP) cells would best be observed in group 1 (placebo). Upon observation of group 1 under original protocol, changes in CEP cells were not significant but there were changes in markers of inflammation, lipids, and HDL protein composition. A modification to the protocol and title were made to reflect this for groups 2 and 3: Hormonal regulation of HDL-C in Men.

DETAILED DESCRIPTION:
We will be administering three drugs: testosterone gel (T), anastrozole, and acyline. We want to see their effects on stem cells and hormone levels in the blood. Acyline suppress luteinizing hormone(LH) and follicle-stimulating hormone(FSH), which are hormones made by the pituitary gland, thus blocking the signal from the brain that causes the testes to make testosterone. Therefore acyline blocks testosterone production. Some men may experience side effects such as hot flashes or irritability from the low levels of T caused by acyline. We are studying whether adding T to acyline will reduce or eliminate these side effects.

Since heart disease is a common problem in men we want to know about the effects of male hormonal contraception on the cardiovascular system. One way to evaluate these risks is to measure the number of progenitor cells and the types of cholesterol in the blood. Progenitor cells are cells that travel in the blood and go to areas of blood vessel injury to help repair the damage amd may help prevent heart attacks and stokes. Some studies suggest that T administration may increase the number of these cells in the blood but other studies have shown that estrogen may be responsible for this effect. In addition, T and estrogen may affect the amount and type of HDL cholesterol in the blood. This is the "good" cholesterol that is thought to protect people from heart attacks and strokes. Therefore, more studies to test the effects of T and estrogen on progenitor cells in the blood and to understand HDL cholesterol in men receiving testosterone are needed.

Acyline is an experimental drug. The FDA allows its use only in research with a small number of volunteers. So far, over 125 men have received acyline. Anastrozole is a drug that blocks the production of estrogen from testosterone. Anastrozole has been given to men safely in the past. Anastrozole is not approved for use in men and is also an experimental drug. Testosterone gel will also be used in this study. It is FDA approved for use in men with low testosterone levels.

ELIGIBILITY:
Inclusion Criteria:

* Males age 18-55 years
* Normal serum total testosterone (300 ng/dl-1000 ng/dl)
* Normal LH and FSH levels
* Taking no regular medications
* Normal baseline serum hematology, chemistry and liver function tests
* Agrees not to donate blood during the study
* Agrees to use a form of contraception during the study
* Subject must be able to comply with all study procedures

Exclusion Criteria:

* Clinically significant screening assessments or other relevant disease, allergy or surgery, as revealed by history, physical examination and/or laboratory assessments, which may limit participation or prevent completion of the study
* History of prostate cancer, breast cancer, or benign prostatic hypertrophy
* Prostate-specific antigen (PSA) > 3.0
* History of regular, chronic testosterone or anabolic steroid use in the past year
* Chronic medical illness, prostate disease, or cardiovascular disease
* History of a bleeding disorder or need for anticoagulation
* Skin condition that might interfere with or be exacerbated by T gel use
* Sitting systolic blood pressure > 180mm Hg or <90 mm Hg or sitting diastolic blood pressure >110 mm Hg or < 60 mm Hg.
* History of clinically significant, untreated sleep apnea
* Participation in another drug-related research study within the past 2 months
* Participating in a regular physical relationship with a pregnant woman
* History of hypersensitivity to any of the study medications (T gel, anastrozole, acyline)
* History of medical or surgical therapy for benign prostatic hypertrophy
* Hematocrit > 55%
* History of drug or alcohol abuse within last 6 months
* Abnormal digital rectal exam at screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Page, MD, PhD, Principal Investigator — University of Washington

REFERENCES:
- [Background] Phillips GB. Is atherosclerotic cardiovascular disease an endocrinological disorder? The estrogen-androgen paradox. J Clin Endocrinol Metab. 2005 May;90(5):2708-11. doi: 10.1210/jc.2004-2011. Epub 2005 Feb 1. PMID 15687329
- [Background] Bebb RA, Anawalt BD, Christensen RB, Paulsen CA, Bremner WJ, Matsumoto AM. Combined administration of levonorgestrel and testosterone induces more rapid and effective suppression of spermatogenesis than testosterone alone: a promising male contraceptive approach. J Clin Endocrinol Metab. 1996 Feb;81(2):757-62. doi: 10.1210/jcem.81.2.8636300.
- [Background] Wu FC, von Eckardstein A. Androgens and coronary artery disease. Endocr Rev. 2003 Apr;24(2):183-217. doi: 10.1210/er.2001-0025. PMID 12700179
- [Background] Keating NL, O'Malley AJ, Smith MR. Diabetes and cardiovascular disease during androgen deprivation therapy for prostate cancer. J Clin Oncol. 2006 Sep 20;24(27):4448-56. doi: 10.1200/JCO.2006.06.2497. PMID 16983113
- [Background] Smith MR. Changes in fat and lean body mass during androgen-deprivation therapy for prostate cancer. Urology. 2004 Apr;63(4):742-5. doi: 10.1016/j.urology.2003.10.063. PMID 15072892
- [Background] Smith MR, Finkelstein JS, McGovern FJ, Zietman AL, Fallon MA, Schoenfeld DA, Kantoff PW. Changes in body composition during androgen deprivation therapy for prostate cancer. J Clin Endocrinol Metab. 2002 Feb;87(2):599-603. doi: 10.1210/jcem.87.2.8299. PMID 11836291
- [Background] Smith MR, Lee H, Nathan DM. Insulin sensitivity during combined androgen blockade for prostate cancer. J Clin Endocrinol Metab. 2006 Apr;91(4):1305-8. doi: 10.1210/jc.2005-2507. Epub 2006 Jan 24. PMID 16434464
- [Background] Braga-Basaria M, Dobs AS, Muller DC, Carducci MA, John M, Egan J, Basaria S. Metabolic syndrome in men with prostate cancer undergoing long-term androgen-deprivation therapy. J Clin Oncol. 2006 Aug 20;24(24):3979-83. doi: 10.1200/JCO.2006.05.9741. PMID 16921050
- [Background] Werner N, Kosiol S, Schiegl T, Ahlers P, Walenta K, Link A, Bohm M, Nickenig G. Circulating endothelial progenitor cells and cardiovascular outcomes. N Engl J Med. 2005 Sep 8;353(10):999-1007. doi: 10.1056/NEJMoa043814. PMID 16148285
- [Background] Werner N, Junk S, Laufs U, Link A, Walenta K, Bohm M, Nickenig G. Intravenous transfusion of endothelial progenitor cells reduces neointima formation after vascular injury. Circ Res. 2003 Jul 25;93(2):e17-24. doi: 10.1161/01.RES.0000083812.30141.74. Epub 2003 Jun 26. PMID 12829619
- [Background] Vasa M, Fichtlscherer S, Aicher A, Adler K, Urbich C, Martin H, Zeiher AM, Dimmeler S. Number and migratory activity of circulating endothelial progenitor cells inversely correlate with risk factors for coronary artery disease. Circ Res. 2001 Jul 6;89(1):E1-7. doi: 10.1161/hh1301.093953. PMID 11440984
- [Background] Dong C, Goldschmidt-Clermont PJ. Endothelial progenitor cells: a promising therapeutic alternative for cardiovascular disease. J Interv Cardiol. 2007 Apr;20(2):93-9. doi: 10.1111/j.1540-8183.2007.00251.x. PMID 17391216
- [Background] Foresta C, Caretta N, Lana A, De Toni L, Biagioli A, Ferlin A, Garolla A. Reduced number of circulating endothelial progenitor cells in hypogonadal men. J Clin Endocrinol Metab. 2006 Nov;91(11):4599-602. doi: 10.1210/jc.2006-0763. Epub 2006 Aug 22. PMID 16926245
- [Background] Foresta C, Zuccarello D, Biagioli A, De Toni L, Prana E, Nicoletti V, Ambrosini G, Ferlin A. Oestrogen stimulates endothelial progenitor cells via oestrogen receptor-alpha. Clin Endocrinol (Oxf). 2007 Oct;67(4):520-5. doi: 10.1111/j.1365-2265.2007.02918.x. Epub 2007 Jun 15. PMID 17573901
- [Background] Foresta C, Zuccarello D, De Toni L, Garolla A, Caretta N, Ferlin A. Androgens stimulate endothelial progenitor cells through an androgen receptor-mediated pathway. Clin Endocrinol (Oxf). 2008 Feb;68(2):284-9. doi: 10.1111/j.1365-2265.2007.03036.x. Epub 2007 Sep 4. PMID 17803706
- [Background] Iwakura A, Luedemann C, Shastry S, Hanley A, Kearney M, Aikawa R, Isner JM, Asahara T, Losordo DW. Estrogen-mediated, endothelial nitric oxide synthase-dependent mobilization of bone marrow-derived endothelial progenitor cells contributes to reendothelialization after arterial injury. Circulation. 2003 Dec 23;108(25):3115-21. doi: 10.1161/01.CIR.0000106906.56972.83. Epub 2003 Dec 15. PMID 14676142
- [Background] Bergt C, Pennathur S, Fu X, Byun J, O'Brien K, McDonald TO, Singh P, Anantharamaiah GM, Chait A, Brunzell J, Geary RL, Oram JF, Heinecke JW. The myeloperoxidase product hypochlorous acid oxidizes HDL in the human artery wall and impairs ABCA1-dependent cholesterol transport. Proc Natl Acad Sci U S A. 2004 Aug 31;101(35):13032-7. doi: 10.1073/pnas.0405292101. Epub 2004 Aug 23. PMID 15326314
- [Background] Leder BZ, LeBlanc KM, Schoenfeld DA, Eastell R, Finkelstein JS. Differential effects of androgens and estrogens on bone turnover in normal men. J Clin Endocrinol Metab. 2003 Jan;88(1):204-10. doi: 10.1210/jc.2002-021036. PMID 12519853
- [Background] Mostaghel EA, Page ST, Lin DW, Fazli L, Coleman IM, True LD, Knudsen B, Hess DL, Nelson CC, Matsumoto AM, Bremner WJ, Gleave ME, Nelson PS. Intraprostatic androgens and androgen-regulated gene expression persist after testosterone suppression: therapeutic implications for castration-resistant prostate cancer. Cancer Res. 2007 May 15;67(10):5033-41. doi: 10.1158/0008-5472.CAN-06-3332. PMID 17510436
- [Background] Page ST, Lin DW, Mostaghel EA, Hess DL, True LD, Amory JK, Nelson PS, Matsumoto AM, Bremner WJ. Persistent intraprostatic androgen concentrations after medical castration in healthy men. J Clin Endocrinol Metab. 2006 Oct;91(10):3850-6. doi: 10.1210/jc.2006-0968. Epub 2006 Aug 1. PMID 16882745
- [Background] Page ST, Plymate SR, Bremner WJ, Matsumoto AM, Hess DL, Lin DW, Amory JK, Nelson PS, Wu JD. Effect of medical castration on CD4+ CD25+ T cells, CD8+ T cell IFN-gamma expression, and NK cells: a physiological role for testosterone and/or its metabolites. Am J Physiol Endocrinol Metab. 2006 May;290(5):E856-63. doi: 10.1152/ajpendo.00484.2005. Epub 2005 Dec 13. PMID 16352669
- [Background] Herbst KL, Coviello AD, Page S, Amory JK, Anawalt BD, Bremner WJ. A single dose of the potent gonadotropin-releasing hormone antagonist acyline suppresses gonadotropins and testosterone for 2 weeks in healthy young men. J Clin Endocrinol Metab. 2004 Dec;89(12):5959-65. doi: 10.1210/jc.2003-032123. PMID 15579744
- [Background] Mauras N, Lima J, Patel D, Rini A, di Salle E, Kwok A, Lippe B. Pharmacokinetics and dose finding of a potent aromatase inhibitor, aromasin (exemestane), in young males. J Clin Endocrinol Metab. 2003 Dec;88(12):5951-6. doi: 10.1210/jc.2003-031279. PMID 14671195
- [Background] Lin EH, Hassan M, Li Y, Zhao H, Nooka A, Sorenson E, Xie K, Champlin R, Wu X, Li D. Elevated circulating endothelial progenitor marker CD133 messenger RNA levels predict colon cancer recurrence. Cancer. 2007 Aug 1;110(3):534-42. doi: 10.1002/cncr.22774. PMID 17594720
- [Background] Hill JM, Zalos G, Halcox JP, Schenke WH, Waclawiw MA, Quyyumi AA, Finkel T. Circulating endothelial progenitor cells, vascular function, and cardiovascular risk. N Engl J Med. 2003 Feb 13;348(7):593-600. doi: 10.1056/NEJMoa022287. PMID 12584367
- [Background] Gonzalo IT, Swerdloff RS, Nelson AL, Clevenger B, Garcia R, Berman N, Wang C. Levonorgestrel implants (Norplant II) for male contraception clinical trials: combination with transdermal and injectable testosterone. J Clin Endocrinol Metab. 2002 Aug;87(8):3562-72. doi: 10.1210/jcem.87.8.8710. PMID 12161475
- [Result] Rubinow KB, Snyder CN, Amory JK, Hoofnagle AN, Page ST. Acute testosterone deprivation reduces insulin sensitivity in men. Clin Endocrinol (Oxf). 2012 Feb;76(2):281-8. doi: 10.1111/j.1365-2265.2011.04189.x. PMID 21797916
- [Result] Rubinow KB, Tang C, Hoofnagle AN, Snyder CN, Amory JK, Heinecke JW, Page ST. Acute sex steroid withdrawal increases cholesterol efflux capacity and HDL-associated clusterin in men. Steroids. 2012 Apr;77(5):454-60. doi: 10.1016/j.steroids.2012.01.002. Epub 2012 Jan 15. PMID 22266332

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited using rosters from prior research studies, newspaper and online advertisements. Recruitment began December 2008 and ended March 2010.
Pre-assignment Details: Before study procedures,2 withdrew consent and 1 was withdrawn by the investigator for missing appointments.4 failed inclusion criteria(1-anemia,1-low testosterone,1-high BMI,1-medications.
  31 men enrolled. 22 men completed.
Groups:
- Group 1: Acyline + Placebo Gel, Placebo Pill: Acyline 300 µg/kg injections Day 0 & 14 + placebo (no active ingredients) transdermal gel daily for 28 days + oral placebo daily for 28 days
- Group 2: Acyline, Testosterone Gel, Placebo Pill: Acyline 300 µg/kg injections Day 0 & 14 + Testosterone gel (Testim) 10g 1% daily for 28 days + oral placebo daily for 28 days
- Group 3: Acyline, Testosterone Gel, Anastrazole Pill: Acyline 300 μg/kg injections Day 0 & 14 + 1% Testosterone gel 10g transdermal daily for 28 days + oral anastrozole 1 mg (Arimidex) daily for 28 days
Period: Overall Study
Arm/Group | Group 1: Acyline + Placebo Gel, Placebo Pill | Group 2: Acyline, Testosterone Gel, Placebo Pill | Group 3: Acyline, Testosterone Gel, Anastrazole Pill
Started | 8 | 8 | 8
Completed | 8 | 6 | 8
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Acyline + Placebo Gel, Placebo Pill | Group 2: Acyline, Testosterone Gel, Placebo Pill | Group 3: Acyline, Testosterone Gel, Anastrazole Pill | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 24
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.5 (10.6) | 24.3 (4.0) | 25.8 (8.4) | 30.0 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 8 | 8 | 8 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 8 | 7 | 7 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 8 | 6 | 7 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (2.5) | 27.1 (3.8) | 23.7 (2.1) | 25.5 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Progenitor Cells
Description: Number of CD33 + CD134+ cells as a percentage of all lymphocytes
Time Frame: Baseline, Day 28
Population: Statistical analyses were limited to changes from baseline within a given group and between-group comparisons were not performed
Measure: Mean (Standard Deviation); unit: percentage of all lymphocytes
Groups:
- Group 1: Acyline + Placebo Gel + Placebo Pill: Group 1: Acyline injections, transdermal placebo gel 10 g/day for 28 days, oral daily placebo pill for 28 days
- Group 2: Acyline + T-gel 10g/Day + Placebo Pill: Acyline SQ inj. Day 0 & 14 + T-gel and placebo pill for 28 days
- Group 3: Acyline + T-gel + Oral Anastrozole 1mg: Acyline SQ inj. Day 0 & 14 + T-gel and anastrozole for 28 days
Arm/Group | Group 1: Acyline + Placebo Gel + Placebo Pill | Group 2: Acyline + T-gel 10g/Day + Placebo Pill | Group 3: Acyline + T-gel + Oral Anastrozole 1mg
Number analyzed (Participants) | 8 | 0 | 0
percentage of all lymphocytes
  Baseline | 0.101 (0.032) |  |
  Day 28 | 0.081 (0.040) |  |
Statistical Analysis 1: Comparison: Group 1: Acyline + Placebo Gel + Placebo Pill; p value for the difference = 0.28; Test type: Superiority or Other; p = 0.28, paired t-test; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [0.005 to 0.035], Standard Deviation 0.0075

2. Secondary Outcome: Follicle Stimulating Hormone (FSH)
Time Frame: Baseline, 28 days
Population: Per protocol, the first 8 subjects were assigned to Group 1. Subsequent subjects were randomly assigned to Group 2 or Group 3.
Measure: Mean (Standard Deviation); unit: IU/L
Groups:
- Group 1: Acyline + Placebo Gel, Placebo Pill: Group 1: Acyline injections, transdermal placebo gel 10 g/day for 28 days, oral daily placebo pill for 28 days
- Group 2: Acyline, Testosterone Gel: Group 2: Acyline injections, transdermal testosterone gel 10 g/day for 28 days, oral daily placebo pill for 28 days
- Group 3: Acyline, Testosterone Gel, Anastrazole Pill: Arm 3: Acyline injections, transdermal testosterone gel 10 g/day for 28 days, oral daily anastrazole pill 1 mg for 28 days
Arm/Group | Group 1: Acyline + Placebo Gel, Placebo Pill | Group 2: Acyline, Testosterone Gel | Group 3: Acyline, Testosterone Gel, Anastrazole Pill
Number analyzed (Participants) | 8 | 6 | 8
IU/L
  Baseline | 4.2 (2.4) | 2.9 (1.3) | 2.5 (0.9)
  Day 28 | 0.42 (0.7) | 0.39 (0.5) | 0.87 (0.8)

3. Secondary Outcome: Luteinizing Hormone Concentration (LH)
Time Frame: Baseline, Day 28
Population: The analysis was per protocol. Following screening, the first 8 subjects were assigned to group I, and subsequent subjects enrolled were randomly assigned to either group 2 or 3.
Measure: Mean (Standard Deviation); unit: IU/L
Groups:
- Group 3: Acyline, Testosterone Gel, Anastrozole: Arm 3: Acyline injections, transdermal testosterone gel 10 g/day for 28 days, oral daily anastrozole pill 1 mg for 28 days.
Arm/Group | Group 1: Acyline + Placebo Gel, Placebo Pill | Group 2: Acyline, Testosterone Gel | Group 3: Acyline, Testosterone Gel, Anastrozole
Number analyzed (Participants) | 8 | 6 | 8
IU/L
  Baseline | 4.3 (2.3) | 4.7 (1.9) | 4.4 (2.2)
  Day 28 | 0.31 (0.2) | 0.69 (1.2) | 1.55 (1.6)

4. Secondary Outcome: Testosterone Concentration
Time Frame: Baseline, Day 28
Population: Per protocol, the first 8 subjects were assigned to group I. Subsequent subjects were randomized to group 2 or group 3.
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- Group 3: Acyline, Testosterone Gel, Anastrozole: Group 3: Acyline injections, transdermal testosterone gel 10 g/day for 28 days, oral daily anastrozole pill 1 mg for 28 days.
Arm/Group | Group 1: Acyline + Placebo Gel, Placebo Pill | Group 2: Acyline, Testosterone Gel | Group 3: Acyline, Testosterone Gel, Anastrozole
Number analyzed (Participants) | 8 | 6 | 8
nmol/L
  Baseline testosterone concentration | 15.4 (3.4) | 16.3 (3.3) | 16.5 (2.6)
  Day 28 testosterone concentration | 0.8 (0.8) | 17.8 (5.5) | 19.0 (7.3)

5. Secondary Outcome: Estradiol Concentration
Time Frame: Baseline, Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pmol/L
Groups:
- Group 3: Acyline, Testosterone Gel, Anastrozole Pill: Group 3: Acyline injections, transdermal testosterone gel 10 g/day for 28 days, oral daily anastrozole pill 1 mg for 28 days.
Arm/Group | Group 1: Acyline + Placebo Gel, Placebo Pill | Group 2: Acyline, Testosterone Gel | Group 3: Acyline, Testosterone Gel, Anastrozole Pill
Number analyzed (Participants) | 8 | 6 | 8
pmol/L
  Baseline | 95.4 (18.2) | 117.8 (28.6) | 96.3 (21.9)
  Day 28 | 31.9 (11.2) | 109.0 (28.8) | 36.5 (14.3)

6. Secondary Outcome: Sex Hormone Binding Globulin (SHBG)
Time Frame: Baseline, Day 28
Population: Per protocol, the first 8 subjects were assigned to Group I. Subsequent subjects were randomly assigned to Group 2 or Group 3.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Group 1: Acyline + Placebo Gel, Placebo Pill | Group 2: Acyline, Testosterone Gel | Group 3: Acyline, Testosterone Gel, Anastrozole Pill
Number analyzed (Participants) | 8 | 6 | 8
nmol/L
  Baseline | 34.9 (17.1) | 23.0 (10.9) | 27.6 (6.3)
  Day 28 | 37.5 (16.4) | 22.1 (10.1) | 25.1 (4.7)

7. Secondary Outcome: Quantitative Insulin Sensitivity Check Index (QUICKI)
Description: QUICKI is a measure of insulin sensitivity calculated using fasting insulin and glucose concentration in a participants blood. Higher QUICKI are associated with decreased insulin resistance and increased insulin sensitivity.
Time Frame: Baseline, Day 28, Day 56
Population: per protocol
Measure: Mean (Standard Deviation); unit: QUICKI index
Groups:
- Group 2: Acyline, Testosterone Gel, Placebo Pill: Group 2: Acyline injections, transdermal testosterone gel 10 g/day for 28 days, oral daily placebo pill for 28 days
- Group 3: Acyline, Testosterone Gel, Oral Anastrozole: Group 3: Acyline injections, transdermal testosterone gel 10 g/day for 28 days, oral daily anastrozole pill 1 mg for 28 days.
Arm/Group | Group 1: Acyline + Placebo Gel, Placebo Pill | Group 2: Acyline, Testosterone Gel, Placebo Pill | Group 3: Acyline, Testosterone Gel, Oral Anastrozole
Number analyzed (Participants) | 8 | 6 | 8
QUICKI index
  Baseline | 0.36 (0.03) | 0.35 (0.02) | 0.36 (0.02)
  Day 28 | 0.34 (0.03) | 0.35 (0.02) | 0.38 (0.02)
  Day 56 | 0.35 (0.03) | 0.35 (0.02) | 0.36 (0.02)

8. Secondary Outcome: Homeostasis Model of Insulin Resistance (HOMA-IR)
Description: HOMA IR is a measure of insulin sensitivity calculated using fasting insulin and glucose concentration in a participants blood. Higher HOMA IR numbers are associated with increased insulin resistance and decreased insulin sensitivity.
Time Frame: Baseline, Day 28, Day 56
Population: per protocol
Measure: Mean (Standard Deviation); unit: HOMA score
Arm/Group | Group 1: Acyline + Placebo Gel, Placebo Pill | Group 2: Acyline, Testosterone Gel, Placebo Pill | Group 3: Acyline, Testosterone Gel, Oral Anastrozole
Number analyzed (Participants) | 8 | 6 | 8
HOMA score
  Baseline | 1.8 (0.9) | 2.0 (0.9) | 1.6 (0.6)
  Day 28 | 2.4 (1.0) | 1.9 (0.9) | 1.4 (0.8)
  Day 56 | 2.2 (0.9) | 1.9 (0.9) | 1.7 (0.8)

9. Secondary Outcome: Fasting Serum Insulin
Time Frame: Baseline, Day 28, Day 56
Population: per protocol
Measure: Mean (Standard Deviation); unit: picomolar
Arm/Group | Group 1: Acyline + Placebo Gel, Placebo Pill | Group 2: Acyline, Testosterone Gel, Placebo Pill | Group 3: Acyline, Testosterone Gel, Oral Anastrozole
Number analyzed (Participants) | 8 | 6 | 8
picomolar
  Baseline | 54 (26) | 65 (28) | 50 (16)
  Day 28 | 69 (25) | 59 (26) | 42 (23)
  Day 56 | 54 (26) | 64 (27) | 50 (16)

10. Secondary Outcome: Fasting Lipid Levels
Time Frame: Baseline, Day 28, Day 56
Population: per protocol
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Group 1: Acyline + Placebo Gel, Placebo Pill | Group 2: Acyline, Testosterone Gel, Placebo Pill | Group 3: Acyline, Testosterone Gel, Oral Anastrozole
Number analyzed (Participants) | 8 | 6 | 8
mmol/L
  Total cholesterol Day 0 | 4.97 (1.1) | 4.48 (0.4) | 4.56 (1.5)
  Total cholesterol Day 28 | 5.44 (1.2) | 4.51 (0.3) | 4.56 (0.9)
  Total cholesterol Day 56 | 4.95 (1.1) | 4.14 (0.6) | 4.27 (1.2)
  LDL choesterol Day 0 | 2.95 (0.8) | 2.77 (0.3) | 2.67 (1.3)
  LDL cholesterol Day 28 | 3.29 (0.7) | 2.80 (0.2) | 2.75 (0.8)
  LDL cholesterol Day 56 | 2.87 (0.5) | 2.49 (0.5) | 2.51 (1.0)
  HDL cholesterol Day 0 | 1.19 (0.2) | 1.32 (0.2) | 1.40 (0.2)
  HDL cholesterol Day 28 | 1.37 (0.2) | 1.32 (0.1) | 1.32 (0.2)
  HDL cholesterol Day 56 | 1.19 (0.2) | 1.32 (0.2) | 1.30 (0.2)
  Triglycerides Day 0 | 1.79 (2.1) | 0.82 (0.2) | 1.08 (0.5)
  Triglycerides Day 28 | 1.73 (1.4) | 0.86 (0.3) | 1.08 (0.4)
  Triglycerides Day 56 | 1.89 (2.3) | 0.80 (0.4) | 1.02 (0.3)

ADVERSE EVENTS:
Time Frame: Dec 2008 - May 2010
Arm/Group | Group 1: Acyline + Placebo Gel, Placebo Pill | Group 2: Acyline, Testosterone Gel, Placebo Pill | Group 3: Acyline, Testosterone Gel, Anastrazole Pill
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 6/8 | 1/6 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Acyline + Placebo Gel, Placebo Pill (N=8) | Group 2: Acyline, Testosterone Gel, Placebo Pill (N=6) | Group 3: Acyline, Testosterone Gel, Anastrazole Pill (N=8)
emotional lability, irritability (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) — This is expected in group 1 subjects (hypogonadal). The group 3 subject with emotional lability also reported skin irritation at the testosterone gel site.
fatigue (Endocrine disorders) | 2 (2) | 1 (1) | 0 (0) — Fatigue is anticipated and consistent with hypogonadal symptoms for Group 1 (placebo gel. The group 2 subject also reported studying late and spending the night in the library during midterm week. Fatigue is described in the consent as a possibility.
hot flashes (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0) — Hot flashes are anticipated and consistent with hypogonadal symptoms for Group 1 (placebo gel). This is described in the consent.
itching at acyline site (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) — The written consent describes itchiness at the site in most men. One (group 2)is not counted here, but is described in "participant flow". Symptoms had resolved on Day 14 but he withdrew consent before the second acyline injection.
lightheadedness, clammy (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) — Mild symptoms occurred two days and were deemed possibly related to the drug. No action or medications were required in this group I (hypogonadal symptoms expected) subject.
low libido (Endocrine disorders) | 4 (4) | 0 (0) | 1 (1) — Low libido is anticipated and consistent with hypogonadal symptoms for Group 1 (placebo gel). This is described in the consent.
skin irritation, gel application site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) — One(group 1) complaint of itchiness;one(group 3) complaint of dry skin at testosterone gel application site. Both subjects were instructed to apply elsewhere; complaints were resolved with no further symptoms at old and new application sites.
itching rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes